CLINICAL TRIAL: NCT00008112
Title: Feasibility Study of the Combination of Radiotherapy, Chemotherapy and Hyperthermia for the Treatment of Stage IIB-III-IVA Cervical Cancer
Brief Title: Cisplatin Combined With Radiation Therapy and Hyperthermia in Treating Patients With Stage II, Stage III, or Stage IV Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DUT-KWF-CKVO-2000-02; CDR0000068376 (Registry Identifier: PDQ (Physician Data Query)); EU-20036
Record Dates: First submitted 2001-01-06; First posted 2003-06-05 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-10

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IIB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Diathermy; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Procedure: hyperthermia treatment
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Combining hyperthermia with radiation therapy and chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin combined with radiation therapy and hyperthermia in treating patients who have stage II, stage III, or stage IV cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of adding cisplatin and locoregional hyperthermia to external beam and intracavity radiotherapy in patients with stage IIB-IVA cervical cancer.
* Determine the acute toxicity of this regimen in these patients.
* Determine the complete response rate of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo external beam radiotherapy (EBRT) once daily 5 days a week for 5 weeks. On 1 day of each week, patients also receive cisplatin IV over 3 hours and hyperthermia over 90 minutes beginning 1-6 hours after completion of EBRT. During week 6, patients receive hyperthermia and cisplatin on the day before the 1 day of intracavity radiotherapy. Treatment continues in the absence of unacceptable toxicity.

Patients are followed at 6-8 weeks, every 3 months for 3 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 6-34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIB-IVA carcinoma of the cervix

  * Adenocarcinoma
  * Squamous cell carcinoma
  * Mixed cell histology
  * No small cell anaplastic histology
* No para-aortic lymph node involvement

  * No indication for para-aortic radiotherapy
* No distant metastases
* No CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 7.0 mmol/L (approximately 11 g/dL)
* Epoetin alfa and/or transfusion allowed

Hepatic:

* Not specified

Renal:

* Glomerular filtration rate at least 60 mL/min

Cardiovascular:

* No myocardial infarction within the past 6 months
* No unstable angina
* No congestive heart failure with expected inability to tolerate fluid load
* No cerebrovascular accident within the past 6 months

Other:

* No pacemaker and/or metal implants
* No active uncontrolled infection
* No compromised immune status
* No psychosis
* No other prior malignancy except nonmelanoma skin cancer
* No mental or other physical inability that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy

Surgery:

* No prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Anneke M. Westermann, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht